CLINICAL TRIAL: NCT01434654
Title: The Efficacy of Neuro-HAART in HIV Infected Individuals
Brief Title: Efficacy of Neuro-HAART in Patients With HIV
Acronym: HANDobs
Status: Terminated | Type: Observational
Why Stopped: Slower than expected recruitment
Sponsor: St Vincent's Hospital, Sydney (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Bruce Brew, Professor, St Vincent's Hospital, Sydney
Other Study IDs: 09/192; COL114560 (Other Grant/Funding Number: VIIV Healthcare)
Record Dates: First submitted 2011-09-12; First posted 2011-09-15 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: HIV
Keywords: HAND; HIV; Neurology; Neurocognitive; Neuro-HAART; HIV Associated Neurocognitive Disorders (HAND)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerbrospinal fluid and bloods
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non Neuro-HAART (low CNS penetrance): Participants will be assessed based on their current Highly Active Antiretroviral Treatment (HAART). A scoring system is utilised to determine if their current treatment has high Central Nervous System (CNS) penetrance or low CNS penetrance. This will determine which study cohort they are allocated to. No treatment adjustments or changes will be made, they will remain on their usual HAART regimen.
- Neuro-HAART (high CNS penetrance): Participants will be assessed based on their current Highly Active Antiretroviral Treatment (HAART). A scoring system is utilised to determine if their current treatment has high Central Nervous System (CNS) penetrance or low CNS penetrance. This will determine which study cohort they are allocated to. No treatment adjustments or changes will be made, they will remain on their usual HAART regimen.

SUMMARY:
Patients infected with Human Immunodeficiency Virus (HIV) are at risk of brain related complications despite the use of highly active antiretroviral therapy (HAART). Such complications are termed HIV neurocognitive disorders (HAND) and comprise a spectrum from asymptomatic neurocognitive impairment (ANI), through mild cognitive impairment (MCI) to severe HIV dementia (HAD).

Prior to HAART approximately 30% of patients with advanced HIV disease had cognitive impairment; with HAART the incidence of HAND has decreased but its prevalence increased. The reasons for the ongoing development of cognitive impairment in HAART treated patients are not clear. They might relate to virus induced brain injury prior to starting HAART, the onset of a separate neurological process, toxicity related to HAART, or ongoing viral infection in the brain.

It is clear that the ability of different antiretroviral drugs to penetrate the brain varies but what is not established is whether these differences between drugs lead to different neurological outcomes. The investigators propose to study HIV infected patients stable on HAART for 12 months; subdividing the groups according to the brain penetrance of their drug combination. Patients would undergo neuropsychological assessment and MRI brain scan at the start of the study and after 12 months.

Differences in neuropsychological tests and MRI would be sought between treatment groups to establish whether HAART with better CNS penetration is associated with better outcome and fewer MRI changes.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive with nadir cluster of differentiation 4 (CD4) count <350 /microlitre (uL)
* Taking HAART with CNS Penetration Effectiveness (CPE) score of either ≤7.0 or ≥7.5 for 1 year or more. Changes in antiretrovirals (ARVs) within the last 12 months are allowed so long as the CPE score does not lead to a change groups
* Plasma HIV viral load <50 copies / mL for preceding 12 months or longer
* Informed consent given by participant or legally appointed guardian

Exclusion Criteria:

* Non-HIV related neurological disorders and active CNS opportunistic infection as assessed by full blood count, electrolytes, creatinine, glucose, liver function tests, cryptococcal antigen, venereal disease reaction level (VDRL), MRI brain scan and cerebrospinal fluid analyses for cell count, protein, glucose, culture, VDRL and cryptococcal antigen.
* Psychiatric disorders on the psychotic axis, current major depression, and current substance use disorder as assessed by the Study Enrolment Questionnaire for Eligibility
* Severe substance use disorders (within 12 months of study entry)
* Active Hepatitis C virus (HCV) (detectable HCV RNA because HCV per se can cause cognitive impairment)
* History of loss of consciousness >1 hour
* Non-proficient in English as assessed by the "English as a second language questionnaire"
* Medications known pharmacologically to interact with ARVs
* Pregnancy as assessed by the urinary pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive participants on HAART who attend outpatient primary care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Brew, MBBS, PhD, Principal Investigator — St Vincent's Hospital, Sydney
Locations (2):
- Australia (2):
  - St Vincent's Hospital, Sydney, New South Wales
  - The Alfred Hospital, Prahran, Victoria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from St Vincent's Hospital and/or referred from tertiary sexual health centres over the period January 2012 to June 2013.
Groups:
- Non Neuro-HAART (Low CNS Penetrance); Neuro-HAART (High CNS Penetrance): Participants will be assessed based on their current Highly Active Antiretroviral Treatment (HAART). A scoring system is utilised to determine if their current treatment has high Central Nervous System (CNS) penetrance or low CNS penetrance. This will determine which study cohort they are randomised to. No treatment adjustments or changes will be made, they will remain on their usual HAART regimen.
Period: Overall Study
Arm/Group | Non Neuro-HAART (Low CNS Penetrance) | Neuro-HAART (High CNS Penetrance)
Started | 7 | 12
Completed | 5 | 12
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data presented reflect baseline demographic and clinical characteristics for participants included in the primary analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non Neuro-HAART (Low CNS Penetrance) | Neuro-HAART (High CNS Penetrance) | Total
Number analyzed (Participants) | 5 | 12 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (7.8) | 55.4 (8.6) | 53.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 12 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 4 | 11 | 15
  Asian | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Australia | 5 | 12 | 17
Education [Mean (Standard Deviation); unit: years] | 14.4 (3.4) | 12.2 (2.7) | 12.8 (2.7)
Premorbid intelligence quotient (IQ) [Mean (Standard Deviation); unit: units on a scale] — Full-scale IQ based on National Adult Reading Test (NART) error score. NART is a test of reading ability that has been extensively validated for use as a proxy measure of pre-morbid intellectual functioning. Full-Scale IQ score is expressed as a Standard Score with Mean=100 and Standard Deviation=15. Possible values range from 69-131. Higher scores indicate better performance.
  units on a scale | 104.2 (18.7) | 102.5 (12.6) | 103.0 (14.1)
Nadir cluster of differentiation 4 (CD4) [Median (Inter-Quartile Range); unit: cells/mm3] | 400 [300.25 to 499.75] | 115 [42.5 to 207.5] | 200 [70 to 330]
Current CD4 [Median (Inter-Quartile Range); unit: cells/mm3] | 943 [752.5 to 1133.5] | 583 [386.25 to 979.75] | 684 [403.25 to 964.75]
HIV-Associated Neurocognitive Disorder (HAND) status [Number; unit: participants]
  Normal/Unimpaired | 1 | 2 | 3
  Asymptomatic Neurocognitive Impairment (ANI) | 2 | 7 | 9
  Mild Neurocognitive Disorder (MND) | 1 | 3 | 4
  HIV-Associated Dementia (HAD) | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Neurocognitive Functioning
Description: Change in overall neurocognitive performance, defined as a global neurocognitive z-score, after a 12-month period of observation, between HIV positive patients taking antiretroviral regimens categorized as being either of high or low CNS penetration. To derive this score, 1) raw scores obtained from a 5-domain brief neurocognitive battery were converted to age-corrected z-scores (M=0, Standard Deviation=1) and 2) the set of individual subtest z-scores were averaged to generate a single composite (global) z-score for each subject. Lower (negative) scores therefore indicate greater levels of cognitive impairment.
Time Frame: Change from baseline Neuropsychological testing at 6 and 12 months
Population: Modified intent-to-treat analysis. All enrolled participants were included aside n=2 low CNS penetrance with baseline data only (1 lost to follow-up, 1 withdrew before 6-months).
Measure: Least Squares Mean (Standard Error); unit: Global neurocognitive z-score
Arm/Group | Non Neuro-HAART (Low CNS Penetrance) | Neuro-HAART (High CNS Penetrance)
Number analyzed (Participants) | 5 | 12
Global neurocognitive z-score
  Baseline | -0.26 (0.27) | -0.80 (0.17)
  6 months | -0.09 (0.27) | -0.63 (0.17)
  12 months | -0.07 (0.27) | -0.61 (0.17)
Statistical Analysis 1: Comparison: Non Neuro-HAART (Low CNS Penetrance) vs Neuro-HAART (High CNS Penetrance); The primary outcome was analysed using a mixed-effect regression model with arm and time as fixed linear effects, arm*time interaction as a non-linear fixed effect and participant as a random effect to account for participant attrition; Test type: Superiority or Other; p = 0.99, Mixed Models Analysis — P-value for arm*time interaction fixed effect; 49 datapoints included from baseline, 6 months, and 12 months visits (low CNS penetrance n=14; high CNS penetrance n=35)

2. Secondary Outcome: Change in MRS Cerebral Metabolite Ratios in Basal Ganglia
Description: Change in major cerebral metabolites in the basal ganglia, as measured by 1H-Magnetic Resonance Spectroscopy (MRS), after a 12 month period of observation. Spectra were acquired on a Phillips Achieva 3T MRI scanner using point-resolved spectroscopy (PRESS) sequence with short echo time (TE). jMRUI/AMARES algorithm was used to process spectra. Metabolite ratios were calculated for the following metabolites: N-acetyl aspartate (NAA), choline (Cho), creatine (Cr), myo-inositol (mIo), in relation to internal water (H20) as standard.
Time Frame: Baseline and 12 months
Population: n=1 participant in high CNS penetrance arm did not return for 12-months follow-up visit. Their baseline data were therefore excluded from analysis.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Non Neuro-HAART (Low CNS Penetrance) | Neuro-HAART (High CNS Penetrance)
Number analyzed (Participants) | 5 | 11
Ratio
  NAA Baseline | 4.14 (0.20) | 4.00 (0.13)
  NAA 12 months | 3.96 (0.20) | 3.99 (0.13)
  Cr Baseline | 3.18 (0.18) | 3.03 (0.12)
  Cr 12 Months | 3.20 (0.18) | 3.27 (0.12)
  Cho Baseline | 1.81 (0.16) | 1.79 (0.11)
  Cho 12 Months | 1.78 (0.16) | 1.72 (0.11)
  mIo Baseline | 1.22 (0.21) | 1.27 (0.14)
  mIo 12 Months | 1.12 (0.21) | 1.18 (0.14)
Statistical Analysis 1: Comparison: Non Neuro-HAART (Low CNS Penetrance) vs Neuro-HAART (High CNS Penetrance); Change in NAA/H20 levels was analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.58, ANOVA
Statistical Analysis 2: Comparison: Non Neuro-HAART (Low CNS Penetrance) vs Neuro-HAART (High CNS Penetrance); Change in Cr/H20 levels was analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.44, ANOVA
Statistical Analysis 3: Comparison: Non Neuro-HAART (Low CNS Penetrance) vs Neuro-HAART (High CNS Penetrance); Change in Cho/H20 levels was analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.86, ANOVA
Statistical Analysis 4: Comparison: Non Neuro-HAART (Low CNS Penetrance) vs Neuro-HAART (High CNS Penetrance); Change in mIo/H20 levels was analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.98, ANOVA

3. Secondary Outcome: Change in MRS Cerebral Metabolite Ratios in Frontal White Matter
Description: Change in major cerebral metabolites in the frontal white matter, as measured by 1H-Magnetic Resonance Spectroscopy (MRS), between baseline and 12-months. Spectra were acquired on a Phillips Achieva 3T MRI scanner using point-resolved spectroscopy (PRESS) sequence with short TE. jMRUI/AMARES algorithm was used to process spectra. Metabolite ratios were calculated for the following metabolites: N-acetyl aspartate (NAA), choline (Cho), creatine (Cr), myo-inositol (mIo), glutamate/glutamine complex (Glx), in relation to internal H20 as standard.
Time Frame: Baseline and 12 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Non Neuro-HAART (Low CNS Penetrance) | Neuro-HAART (High CNS Penetrance)
Number analyzed (Participants) | 5 | 11
Ratio
  NAA Baseline | 4.39 (0.22) | 4.38 (0.15)
  NAA 12 Months | 4.74 (0.22) | 4.32 (0.15)
  Cr Baseline | 2.77 (0.19) | 3.09 (0.12)
  Cr 12 Months | 3.29 (0.19) | 3.16 (0.12)
  Cho Baseline | 2.25 (0.13) | 2.33 (0.09)
  Cho 12 Months | 2.50 (0.13) | 2.31 (0.08)
  mIo Baseline | 1.06 (0.09) | 1.05 (0.06)
  mIo 12 Months | 1.19 (0.09) | 1.23 (0.06)
  Glx Baseline | 2.26 (0.16) | 2.13 (0.11)
  Glx 12 Months | 2.13 (0.19) | 1.96 (0.11)
Statistical Analysis 1: Comparison: Non Neuro-HAART (Low CNS Penetrance) vs Neuro-HAART (High CNS Penetrance); Change in NAA/H20 levels were analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.16, ANOVA
Statistical Analysis 2: Comparison: Non Neuro-HAART (Low CNS Penetrance) vs Neuro-HAART (High CNS Penetrance); Change in Cr/H20 levels were analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.09, ANOVA
Statistical Analysis 3: Comparison: Non Neuro-HAART (Low CNS Penetrance) vs Neuro-HAART (High CNS Penetrance); Change in Cho/H20 levels were analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.06, ANOVA
Statistical Analysis 4: Comparison: Non Neuro-HAART (Low CNS Penetrance) vs Neuro-HAART (High CNS Penetrance); Change in mIo/H20 levels were analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.68, ANOVA
Statistical Analysis 5: Comparison: Non Neuro-HAART (Low CNS Penetrance) vs Neuro-HAART (High CNS Penetrance); Change in Glx/H20 levels were analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.58, ANOVA

4. Secondary Outcome: Cerebrospinal Fluid
Description: To measure plateaux CSF ARV concentrations. This will identify the proportion of patients achieving levels of specific ARVs capable of inhibiting 95% of in vitro viral replication (IC95).
Time Frame: Baseline to 12 Months
Population: Data presented for n=5 participants with detectable CSF ARV concentrations who had lumbar puncture at Baseline and 12 months. The pre-specified analysis was not conducted as nevirapine, raltegravir, and darunavir were the only ARVs detected in CSF, and of these, only nevirapine was detected above the minimum threshold (set at >50 ug/L).
Measure: Mean (Standard Error); unit: ug/L
Arm/Group | Non Neuro-HAART (Low CNS Penetrance) | Neuro-HAART (High CNS Penetrance)
Number analyzed (Participants) | 1 | 4
ug/L
  Nevirapine Baseline | NA (NA) — No participants in this study arm had detectable nevirapine CSF concentrations at baseline. Therefore no data available to report. | 1161.5 (101.5)
  Nevirapine 12 months | NA (NA) — No participants in this study arm had detectable nevirapine CSF concentrations at 12 months. Therefore no data available to report. | 1445 (234)
  Raltegravir Baseline | 38 (NA) — n=1 participant in this study arm had detectable raltegravir CSF concentrations at baseline. Therefore SE not applicable. | 39 (NA) — n=1 participant in this study arm had detectable raltegravir CSF concentrations at baseline. Therefore SE not applicable.
  Raltegravir 12 months | 32 (NA) — n=1 participant in this study arm had detectable raltegravir CSF concentrations at 12 months. Therefore SE not applicable. | NA (NA) — No participants in this study arm had detectable raltegravir CSF concentrations at 12 months. Therefore no data available to report.
  Darunavir Baseline | 46 (NA) — n=1 participant in this study arm had detectable darunavir CSF concentrations at baseline. Therefore SE not applicable. | 39 (NA) — n=1 participant in this study arm had detectable darunavir CSF concentrations at baseline. Therefore SE not applicable.
  Darunavir 12 months | NA (NA) — No participants in this study arm had detectable darunavir CSF concentrations at 12 months. Therefore no data available to report. | 50 (NA) — n=1 participant in this study arm had detectable darunavir CSF concentrations at 12 months. Therefore SE not applicable.

ADVERSE EVENTS:
Time Frame: Baseline to 12 Months
Arm/Group | Non Neuro-HAART (Low CNS Penetrance) | Neuro-HAART (High CNS Penetrance)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/12
Other Adverse Events (participants affected / at risk) | 2/7 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Neuro-HAART (Low CNS Penetrance) (N=7) | Neuro-HAART (High CNS Penetrance) (N=12)
Post-lumbar puncture headache (Investigations) | 1 (1) | 1 (1)
Laser eye surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Kidney stones and stent insertion (Renal and urinary disorders) | 1 (1) | 0 (0)
Rash and excema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin biopsy (Investigations) | 0 (0) | 1 (1)
Basal cell carcinoma removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Lower than expected participant recruitment rate and early termination led to a small sample size and underpowered statistical analyses

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No